CLINICAL TRIAL: NCT01783964
Title: An Open-Label, Single-Dose Study Designed to Assess the Mass Balance Recovery of an Intravenous Microdose of [14C]-Elacytarabine in Healthy Male Subjects
Brief Title: Elacytarabine Mass Balance Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clavis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CP4055-110
Record Dates: First submitted 2013-02-01; First posted 2013-02-05 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Not Applicable as This is a Mass Balance/Pharmacokinetic Study Performed in Healthy Subjects
Keywords: Elacytarabine; pharmacokinetic; Microdose; Mass Balance Recovery
MeSH Terms: interventions — 5'-oleoyl cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]-Elacytarabine Microdose (Experimental): intravenous (IV) administration of one dose of elacytarabine
  Interventions: Drug: [14C]-Elacytarabine

INTERVENTIONS:
Drug: [14C]-Elacytarabine — Single intravenous administration
  Other Names: elacytarabine

SUMMARY:
This study is performed to measure the quantity of i.v. applied elacytarabine that leave the body, by which route and how fast.

DETAILED DESCRIPTION:
This is a single centre, open-label, non-randomised single dose study in healthy male subjects. Each subject will receive a single 15 min IV administration of 14C labelled elacytarabine.

In this study, at least 6 subjects will be dosed in order to obtain data in 4 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males 2. Age 50 to 65 years of age 4. Must be willing and able to communicate and participate in the whole study 5. Must provide written informed consent 6. Must agree to use an adequate method of contraception

Exclusion Criteria:

1. Participation in a clinical research study within the previous 3 months
2. Subjects who are study site employees, or immediate family members of a study site or sponsor employee
3. Subjects who have previously been enrolled in this study or in any other elacytarabine study
4. History of any drug or alcohol abuse in the past 2 years

7. Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999, shall participate in the study 8. Subjects who do not have suitable veins for multiple venepunctures and IV administration as assessed by the investigator at screening 9. Clinically significant abnormal biochemistry, haematology or urinalysis as judged by the investigator 10. Positive drugs of abuse test result 11. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results 12. History of cardiovascular, renal, hepatic, chronic respiratory or gastrointestinal disease as judged by the investigator 13. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients 14. Presence or history of allergy requiring treatment. Hayfever is allowed unless it is active 15. Donation or loss of greater than 400 mL of blood within the previous 3 months 16. Subjects who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies in the 14 days before IMP administration 17. Failure to satisfy the investigator of fitness to participate for any other reason

Ages: 50 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
mass balance of elacytarabine after i.v. dosing | Two weeks after administration
  Blood samples for determination of total radioactivity in whole blood will be withdrawn at pre dose, 3 h, 9 h, 24 h, 48 h, 72 h, 96 h, 120 h, 144 h and 168 h post-dose and at admission on Days 10 and 14.
  No pharmacokinetic parameter estimations will be performed on the whole blood total radioactivity data.
  Urine samples will be collected daily for Days 1 to 7 (i.e., ending on the morning of Day 8) and for a 24 h period on Days 10 and 14. On Day 1, urine collections will be pre dose, 0 to 6, 6 to 12 and 12 to 24 h post dose. Thereafter collections will be for 24 h periods Faecal samples will be collected pre-dose and daily for Days 1 to 7 (i.e., ending on the morning of Day 8), 10 and 14 (wherever possible)

SECONDARY OUTCOMES:
To provide safety and tolerability information for elacytarabine given as a microdose | Two weeks after administration
  * Clinical chemistry, haematology and urinalysis assessments will be performed at screening, pre-dose, 168 h post-dose and at admission on Day 14
  * Electrocardiograms (ECG) will be performed at screening, admission on Day -1, and at 4 h and 168 h post-dose.
  * Vital signs (heart rate and blood pressure) will be performed at screening, admission on Day -1, pre-dose, at the end of the infusion and at 1 h, 4 h, 24 h and 168 h post-dose.
  * Temperature will be performed on admission on Day -1 and pre-dose.
  * Physical examinations will be performed at screening.
  * Drugs of abuse tests, and alcohol and carbon monoxide breath tests will be performed at screening and at admission on Day -1.
  * Subjects will be tested for hepatitis B, hepatitis C and human immunodeficiency virus at screening.
  * Adverse events (AEs) will be monitored throughout the study. Any AEs that are ongoing at discharge from the study on Day 15 will be followed up until stable or resolution

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Clinical, Ruddington, Nottngham, United Kingdom